CLINICAL TRIAL: NCT00631423
Title: Clinical Course and Prognosis of Patients With Vena Cava Inferior Thrombosis
Brief Title: Evaluation of Patients With Vena Cava Inferior Thrombosis
Status: Completed | Type: Observational
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Responsible Party: Principal Investigator, Birgit Linnemann, M.D., Johann Wolfgang Goethe University Hospital
Other Study IDs: E 102/7
Record Dates: First submitted 2008-02-27; First posted 2008-03-07 (Estimated); Last update posted 2015-04-15 (Estimated); Status verified 2015-04

CONDITIONS: Inferior Vena Cava Thrombosis; Venous Thromboembolism
MeSH Terms: conditions — Venous Thromboembolism

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Patients with vena cava inferior thrombosis
- 2: Patients with isolated lower-extremity DVT matched for gender and age

SUMMARY:
The purpose of the study is to evaluate patients with inferior vena cava (IVC)thrombosis in terms of etiology, clinical course and prognosis during long-term follow-up. Patients with isolated lower extremity DVT, matched for age and gender, serve as controls.

DETAILED DESCRIPTION:
All Patients are assessed using a standardized questionnaire and details concerning VTE risk factors, concomitant disease, medical conditions, diagnosis and therapy of IVC thrombosis were registered. A blood sample is taken to test for inherited and acquired thrombophilia. In addition, duplex ultrasound examination and digital photoplethysmograph are performed to assess postthrombotic syndrome.

ELIGIBILITY:
Inclusion Criteria:

* age 18-90 years

Exclusion Criteria:

* none

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with venous thrombosis involving the inferior cava inferior obtained from the Main-Isar-Thrombosis registry in which all patients seen for venous thromboembolism in our department are registered
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2007-07; Primary Completion 2014-04 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Recurrent venous thromboembolism | 6, 12, 24 and 60 months

SECONDARY OUTCOMES:
All-cause mortality | 6, 12, 24 and 60 months
Post-thrombotic syndrome | 24 and 60 months

CONTACTS AND LOCATIONS:
Overall Officials: Birgit Linnemann, MD, Principal Investigator — Division of Vascular Medicine, Department of Internal Medicine, J.W.Goethe University Hospital Frankfurt/Main, Germany
Locations (1):
- Division of Vascular Medicine, Department of Internal Medicine, J.W.Goethe University Hospital Frankfurt, Frankfurt am Main, Hesse, Germany